CLINICAL TRIAL: NCT05525078
Title: E-cigarettes as Harm Reduction Tools in Smokers Who Fail to Quit With Traditional Methods
Brief Title: Quit or Switch: E-cigarette Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Tracy Smith, Assistant Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO#00118102
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — Electronic Nicotine Delivery Systems; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Switch Group (Experimental): Participants in the Switch group will receive a 5-week supply of e-cigarettes.
  Interventions: Behavioral: e-cigarette
- Meds Group (Active Comparator): Participants in the Meds Group will receive a 5-week supply of combination nicotine replacement therapy (transdermal nicotine patch and short-acting nicotine lozenge).
  Interventions: Other: Nicotine patch, Nicotine lozenge

INTERVENTIONS:
Behavioral: e-cigarette — Participants will select a Target Switch on which they will stop smoking cigarettes and switch entirely to the e-cigarette product.
  Arms: Switch Group
Other: Nicotine patch, Nicotine lozenge — Participants will select a Target Quit Date on which they will stop smoking, using the patches and lozenges provided.
  Arms: Meds Group

SUMMARY:
The majority of smokers try to quit each year, and the majority of quit attempts fail, even when the most effective FDA-approved pharmacotherapies are used. Non-combustible tobacco products emit fewer harmful chemicals than cigarettes, and thus for smokers who cannot quit smoking, switching completely to a less harmful product is likely to improve their risk of cancer and other deleterious health outcomes. E-cigarettes, the most commonly used non-cigarette tobacco product, have been shown to deliver sufficient nicotine, be appealing to smokers, and reduce cigarette smoking when provided to smokers to use ad libitum. For smokers who have failed to quit with traditional methods, trying to switch to a less harmful product may be more likely to help them stop smoking than trying to quit using tobacco altogether repeatedly with pharmacotherapy. The proposed trial evaluates the potential of e-cigarettes to serve as harm reduction tools for current smokers who have already tried, and failed, to quit with traditional methods. Current smokers who failed to quit with FDA-approved pharmacotherapy within the past year (N=30) will be randomly assigned to either 1) switch completely to e-cigarettes (Switch Group, n=20), or 2) try to quit again using pharmacotherapy (Meds Group, n=10). Thus, our design is strengthened by a strong active control group. Participants will select a Target Switch / Quit Date on which they will stop smoking. Participants in the Switch group will receive a 5-week supply of JUUL e-cigarettes, the most popular e-cigarette currently available. Participants in the Meds Group will receive a 5-week supply of combination nicotine replacement therapy (transdermal nicotine patch and short-acting nicotine lozenge). Participants will use 1-week of their tobacco product or medication ad libitum while continuing to smoke in advance of their Target Switch / Quit Date, and 4-weeks as instructed following a Target Switch or Quit Date. Behavioral outcomes of interest include smoking reduction > 50% and biochemically-confirmed abstinence from cigarette smoking at 4-weeks. The proposed trial addresses a highly significant research question using a rigorous design and is supported by a strong investigative team.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years old
2. Smoking at least 5 cigarettes per day for 1 year
3. A quit attempt using an FDA-approved pharmacotherapy in the past year that resulted in abstinence of at least 24 hours
4. Intention to quit smoking within the next month
5. Access to daily e-mail or a smartphone that receives text messages

Exclusion Criteria:

1. use of non-cigarette tobacco products in the past 30 days
2. current use of pharmacotherapy for smoking cessation
3. pregnant, breastfeeding, or trying to become pregnant
4. household member currently enrolled in the study
5. contraindicated for NRT
6. planning to move out of the area within the next 6 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Switch Group | Meds Group
Started | 20 | 10
Completed | 18 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Switch Group | Meds Group | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (12.8) | 49.6 (10.3) | 50.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 17 | 9 | 26
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Report Daily Use of E-cigarettes or NRT and no Cigarette Use
Description: daily use of e-cigarette or NRT instead of cigarettes
Time Frame: day 0 through day 35
Reporting Status: Not Posted

2. Primary Outcome: Percentage of Participants Who Have Biochemically-confirmed Abstinence From Cigarette Smoking at Week 4
Description: Self reported point prevalence abstinence from cigarettes and expired carbon monoxide < 6 ppm
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Switch Group | Meds Group
Number analyzed (Participants) | 20 | 10
Participants | 7 | 1

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Switch Group | Meds Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/10
Other Adverse Events (participants affected / at risk) | 8/20 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch Group (N=20) | Meds Group (N=10)
Suicidal Thoughts (Psychiatric disorders) | 0 (0) | 1 (1) — Severe suicidal thoughts
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Switch Group (N=20) | Meds Group (N=10)
Burning, mucus, or irritation in the throat/sinuses (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Changes in taste/dry mouth (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Insomnia or dream abnormalities (Nervous system disorders) | 0 (0) | 4 (4)
Nausea, flatulence, or stomachache (Gastrointestinal disorders) | 0 (0) | 1 (2)
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Throat or mouth irritation/ulcers (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Vertigo or Dizziness (Ear and labyrinth disorders) | 2 (2) | 0 (0)
headaches (Cardiac disorders) | 1 (1) | 4 (4)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1)
short of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
brochitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
increased mucus / phlegm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/78/NCT05525078/Prot_SAP_002.pdf
  • Informed Consent Form (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT05525078/ICF_001.pdf